CLINICAL TRIAL: NCT06605911
Title: Assessment of the Efficacy of Topical Applied Curcumin 1% as Alternative or Complementary to Triamcinolone Acetonate in Treatment of Oral Lichen Planus(Randomise Control Trial)
Brief Title: Assessment of the Efficacy of Topical Curcumin in Treatment of Oral Lichen Planus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shaymaa Hussein Rafat Kotb (Other)
Responsible Party: Sponsor-Investigator, Shaymaa Hussein Rafat Kotb, Assistant lecturer of Oral Medicine ,periodontology ,oral Diagnosis & Dental Radiology ,Sphinx university, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AUAREC20240004-15
Record Dates: First submitted 2024-09-10; First posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Oral Lichen Planus
Keywords: oral lichen planus; Immune mediated condition; Topical Curcumin; Interlukin 6; ELIZA; Topical triamcinolone acetonide
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Triamcinolone Acetonide; Curcumin

STUDY DESIGN:
Intervention Model Description: thirty patients with oral lichen planus were divided into three groups, 10 patients each: Group A: ten patients with OLP were received topical triamcinolone acetonide. Group B: ten patients with OLP were received topical curcumin. Group C: ten patients with oral lichen planus were received topical triamcinolone acetonide combiend with topical curcumin. For six weeks. Each patient was examined at baseline, 2, weeks and 1 and 3months of therapy. Pain was scored using the visual analogue scale. Salivary level of interleukin 1 were estimated at baseline, 1 and3 months' evaluation periods.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Topical triamcinolone acetonide (Experimental): Group I
  Interventions: Drug: topical triamcinolone acetonide
- Topical curcumin (Experimental): Group II
  Interventions: Drug: Topical Curcumin
- Topical triamcinolone acetonide combiend with topical curcumin (Active Comparator): Group III
  Interventions: Drug: topical triamcinolone acetonide combiend with topical curcumin

INTERVENTIONS:
Drug: topical triamcinolone acetonide — ten patients with OLP were received topical triamcinolone acetonide four times per day for six weeks
  Other Names: Group I
  Arms: Topical triamcinolone acetonide
Drug: Topical Curcumin — Ten patients with OLP received topical curcumin four times per day for six weeks.
  Other Names: Group II
  Arms: Topical curcumin
Drug: topical triamcinolone acetonide combiend with topical curcumin — Ten patients with OLP received a combination of topical triamcinolone acetonide and topical curcumin four times per day for six weeks.
  Other Names: Group III
  Arms: Topical triamcinolone acetonide combiend with topical curcumin

SUMMARY:
to evaluate the therapeutic impact of curcumin as Alternative or Complementary to Triamcinolone Acetonate in Treatment of Oral Lichen Planus.

DETAILED DESCRIPTION:
Background: Oral lichen planus (OLP) is a chronic inflammatory disorder affecting the mucous membranes, believed to be an immune-mediated condition. Its persisting nature can lead to extended discomfort for those affected. The primary symptoms are pain and a burning sensation, with a potential risk of malignancy if not properly managed, necessitating lifelong clinical monitoring. Presently, OLP is considered a significant challenge due to the absence of a definitive cure.

Patients & patients: Thirty patients with oral lichen planus were divided into three groups, 10 patients each: Group A: ten patients with OLP were received topical triamcinolone acetonide. Group B: ten patients with OLP were received topical curcumin. Group C: ten patients with oral lichen planus were received topical triamcinolone acetonide combiend with topical curcumin. For six weeks. Each patient was examined at baseline,1 and 3months of therapy. Pain was scored using the visual analogue scale. Salivary level of interleukin 1 were estimated at baseline,1and 3 months' evaluation periods.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of OLP

Exclusion Criteria:

* Any systemic autoimmune disease
* Any current use of anticoagulant or antiplatelet agents (curcumin has inhibitory effects on platelet aggregations).
* Any topical, local or systemic corticosteroids therapy during the past 3 months.
* lichenoid reaction from medications.
* Pregnant or lactation women.
* smokers

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Assess Visual Analog Scale (VAS) of OLP lesion | baseline ,1 ,3 months
  Qualitative.P-value >0.05: Non significant(NS); P-value <0.05: Significant(S); P-value< 0.01: highly significant(HS)
Assess Oral Disease Severity Score | at base line ,after 1,3 months
  Qualitative.P-value >0.05: Non significant(NS); P-value <0.05: Significant(S); P-value< 0.01: highly significant(HS)

SECONDARY OUTCOMES:
Biochemical analysis of salivary interlukin 6 level using (ELISA) | baseline ,1 ,3 months
  Quantity

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed F Edrees, prof, Study Director — Al-AzharU
Locations (1):
- Al-Azhar university, Asyut, Ass, Egypt

REFERENCES:
- See also: Orchid — https://orcid.org/my-orcid?orcid=0000-0002-8404-438X